CLINICAL TRIAL: NCT00919867
Title: A Phase 1, Open-label, Randomized, Three-period Crossover Drug Interaction Study Evaluating the Pharmacokinetic Profiles of SPD503 and VYVANSE, Administered Alone and in Combination in Healthy Adult Volunteers
Brief Title: A Drug Interaction Study of SPD503 and Vyvanse Administered Alone and In Combination in Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SPD503-115
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Results first posted 2010-08-02 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Healthy
Keywords: Normal, healthy volunteers (for this Phase 1 study)
MeSH Terms: interventions — Guanfacine; Lisdexamfetamine Dimesylate

ARMS (3):
- A: SPD503 (4mg) (Active Comparator)
  Interventions: Drug: SPD503
- B: VYVANSE (50mg) (Active Comparator)
  Interventions: Drug: VYVANSE
- C: SPD503 (4mg) + VYVANSE (50mg) (Active Comparator)
  Interventions: Drug: SPD503 and VYVANSE

INTERVENTIONS:
Drug: SPD503 — SPD503 extended-release 4mg orally administered tablets. There are 3 dosing periods in the study. Subjects will receive one dosing regimen (arm) as a single oral dose on the first day of each dosing period. The order in which the subjects receive each arm (regimen) is randomly assigned. There is a 7-day break between each dosing period in which no medication is taken.
  Other Names: guanfacine hydrochloride
  Arms: A: SPD503 (4mg)
Drug: VYVANSE — VYVANSE 50mg orally administered capsules. There are 3 dosing periods in the study. Subjects will receive one dosing regimen (arm) as a single oral dose on the first day of each dosing period. The order in which the subjects receive each arm (regimen) is randomly assigned. There is a 7-day break between each dosing period in which no medication is taken.
  Other Names: lisdexamfatamine dimesylate (LDX)
  Arms: B: VYVANSE (50mg)
Drug: SPD503 and VYVANSE — SPD503 4mg tablets + VYVANSE 50mg capsules orally administered together. There are 3 dosing periods in the study. Subjects will receive one dosing regimen (arm) as a single oral dose on the first day of each dosing period. The order in which the subjects receive each arm (regimen) is randomly assigned. There is a 7-day break between each dosing period in which no medication is taken.
  Arms: C: SPD503 (4mg) + VYVANSE (50mg)

SUMMARY:
Drug-drug interaction study; to examine the pharmacokinetics of SPD503 and VYVANSE (lisdexamfetamine dimesylate) when given alone, and in combination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be normal healthy adult volunteers (with no significant abnormalities in medical history, physical exam, vital signs or lab evaluations at screening) in order to be eligible to participate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-06-24 (Actual); Primary Completion 2009-07-30 (Actual); Study Completion 2009-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Advanced Biomedical Research, Inc., Hackensack, New Jersey, United States

REFERENCES:
- [Result] Roesch B, Corcoran ME, Fetterolf J, Haffey M, Martin P, Preston P, Purkayastha J, Wang P, Ermer J. Pharmacokinetics of coadministered guanfacine extended release and lisdexamfetamine dimesylate. Drugs R D. 2013 Jun;13(2):119-28. doi: 10.1007/s40268-013-0014-8. PMID 23615868

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study consists of 3 treatment periods performed in 6 dosing sequences: SPD503 (extended-release guanfacine HCl) single 4 mg dose, Vyvanse (lisdexamfatamine dimesylate ) single 50 mg dose, and SPD503 (single 4 mg dose) + Vyvanse (single 50 mg dose) coadministered. There is a washout period between each treatment period.
Groups:
- SPD503 First, Then Vyvanse, Then SPD503 + Vyvanse: SPD503 single 4 mg dose in first intervention, washout, Vyvanse single 50 mg dose in second intervention, washout, SPD503 (single 4 mg dose) + Vyvanse (single 50 mg dose) coadministered in third intervention
- SPD503 First, Then SPD503 + Vyvanse, Then Vyvanse: SPD503 single 4 mg dose in first intervention, washout, SPD503 (single 4 mg dose) + Vyvanse (single 50 mg dose) coadministered in second intervention, washout, Vyvanse single 50 mg dose in third intervention
- Vyvanse First, Then SPD503, Then SPD503 + Vyvanse: Vyvanse single 50 mg dose in first intervention, washout, SPD503 single 4 mg dose in second intervention, washout, SPD503 (single 4 mg dose) + Vyvanse (single 50 mg dose) coadministered in third intervention
- Vyvanse First, Then SPD503 + Vyvanse, Then SPD503: Vyvanse single 50 mg dose in first intervention, washout, SPD503 (single 4 mg dose) + Vyvanse (single 50 mg dose) coadministered in second intervention, washout, SPD503 single 4 mg dose in third intervention
- SPD503 + Vyvanse First, Then SPD503, Then Vyvanse: SPD503 (single 4 mg dose) + Vyvanse (single 50 mg dose) coadministered in first intervention, washout, SPD503 single 4 mg dose in second intervention, washout, Vyvanse single 50 mg dose in third intervention
- SPD503 + Vyvanse, Then Vyvanse, Then SPD503: SPD503 (single 4 mg dose) + Vyvanse (single 50 mg dose) coadministered in first intervention, washout, Vyvanse single 50 mg dose in second intervention, washout, SPD503 single 4 mg dose in third intervention
Period: First Intervention
Arm/Group | SPD503 First, Then Vyvanse, Then SPD503 + Vyvanse | SPD503 First, Then SPD503 + Vyvanse, Then Vyvanse | Vyvanse First, Then SPD503, Then SPD503 + Vyvanse | Vyvanse First, Then SPD503 + Vyvanse, Then SPD503 | SPD503 + Vyvanse First, Then SPD503, Then Vyvanse | SPD503 + Vyvanse, Then Vyvanse, Then SPD503
Started | 7 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 6 | 7 | 7 | 6
Not Completed | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1
Period: Washout
Arm/Group | SPD503 First, Then Vyvanse, Then SPD503 + Vyvanse | SPD503 First, Then SPD503 + Vyvanse, Then Vyvanse | Vyvanse First, Then SPD503, Then SPD503 + Vyvanse | Vyvanse First, Then SPD503 + Vyvanse, Then SPD503 | SPD503 + Vyvanse First, Then SPD503, Then Vyvanse | SPD503 + Vyvanse, Then Vyvanse, Then SPD503
Started | 7 | 7 | 6 | 7 | 7 | 6
Completed | 7 | 7 | 6 | 7 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | SPD503 First, Then Vyvanse, Then SPD503 + Vyvanse | SPD503 First, Then SPD503 + Vyvanse, Then Vyvanse | Vyvanse First, Then SPD503, Then SPD503 + Vyvanse | Vyvanse First, Then SPD503 + Vyvanse, Then SPD503 | SPD503 + Vyvanse First, Then SPD503, Then Vyvanse | SPD503 + Vyvanse, Then Vyvanse, Then SPD503
Started | 7 | 7 | 6 | 7 | 7 | 6
Completed | 7 | 7 | 6 | 7 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | SPD503 First, Then Vyvanse, Then SPD503 + Vyvanse | SPD503 First, Then SPD503 + Vyvanse, Then Vyvanse | Vyvanse First, Then SPD503, Then SPD503 + Vyvanse | Vyvanse First, Then SPD503 + Vyvanse, Then SPD503 | SPD503 + Vyvanse First, Then SPD503, Then Vyvanse | SPD503 + Vyvanse, Then Vyvanse, Then SPD503
Started | 7 | 7 | 6 | 7 | 7 | 6
Completed | 7 | 7 | 6 | 7 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | SPD503 First, Then Vyvanse, Then SPD503 + Vyvanse | SPD503 First, Then SPD503 + Vyvanse, Then Vyvanse | Vyvanse First, Then SPD503, Then SPD503 + Vyvanse | Vyvanse First, Then SPD503 + Vyvanse, Then SPD503 | SPD503 + Vyvanse First, Then SPD503, Then Vyvanse | SPD503 + Vyvanse, Then Vyvanse, Then SPD503
Started | 7 | 7 | 6 | 7 | 7 | 6
Completed | 7 | 7 | 6 | 7 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SPD503 First, Then Vyvanse, Then SPD503 + Vyvanse | SPD503 First, Then SPD503 + Vyvanse, Then Vyvanse | Vyvanse First, Then SPD503, Then SPD503 + Vyvanse | Vyvanse First, Then SPD503 + Vyvanse, Then SPD503 | SPD503 + Vyvanse First, Then SPD503, Then Vyvanse | SPD503 + Vyvanse, Then Vyvanse, Then SPD503 | Total
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 7 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 7 | 7 | 7 | 7 | 42
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (6.20) | 28.7 (8.44) | 34.6 (10.18) | 26.0 (5.29) | 31.9 (8.19) | 31.1 (4.18) | 30.5 (7.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 2 | 2 | 1 | 9
  Male | 6 | 6 | 5 | 5 | 5 | 6 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 7 | 7 | 7 | 7 | 42

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Guanfacine
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 30, 48 and 72 hours post-dose
Population: Pharmacokinetic Population (PKP) consists of all subjects in the Safety Population who had evaluable concentration-time profiles for guanfacine or d-amphetamine. The Safety Population consists of all subjects who received at least 1 dose of study drug and had at least 1 post-dose safety assessment.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- SPD503 Alone: Single 4 mg dose of extended-release Guanfacine HCl
- SPD503 + Vyvanse: SPD503 (single 4 mg dose) + Vyvanse (single 50 mg dose) coadministered
Arm/Group | SPD503 Alone | SPD503 + Vyvanse
Number analyzed (Participants) | 40 | 41
ng/ml | 2.55 (1.03) | 2.97 (0.98)

2. Primary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUC) of Guanfacine
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 30, 48 and 72 hours post-dose
Population: PKP
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | SPD503 Alone | SPD503 + Vyvanse
Number analyzed (Participants) | 37 | 39
ng*h/ml | 104.9 (34.7) | 112.8 (35.7)

3. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) of Guanfacine
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 30, 48 and 72 hours post-dose
Population: PKP
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | SPD503 Alone | SPD503 + Vyvanse
Number analyzed (Participants) | 40 | 41
hours | 8.6 (7.7) | 7.9 (5.0)

4. Primary Outcome: Time of Plasma Half-Life(T 1/2) of Guanfacine
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 30, 48 and 72 hours post-dose
Population: PKP
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | SPD503 Alone | SPD503 + Vyvanse
Number analyzed (Participants) | 37 | 39
hours | 23.5 (10.2) | 21.4 (8.2)

5. Primary Outcome: Cmax of d-Amphetamine
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 30, 48 and 72 hours post-dose
Population: PKP
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Vyvanse Alone: Single 50 mg dose
Arm/Group | Vyvanse Alone | SPD503 + Vyvanse
Number analyzed (Participants) | 41 | 41
ng/ml | 36.48 (7.13) | 36.50 (6.00)

6. Primary Outcome: AUC of d-Amphetamine
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 30, 48 and 72 hours post-dose
Population: PKP
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Vyvanse Alone | SPD503 + Vyvanse
Number analyzed (Participants) | 41 | 41
ng*h/ml | 686.9 (159.8) | 708.4 (137.8)

7. Primary Outcome: Tmax of d-Amphetamine
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 30, 48 and 72 hours post-dose
Population: PKP
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Vyvanse Alone | SPD503 + Vyvanse
Number analyzed (Participants) | 41 | 41
hours | 4.2 (1.1) | 3.9 (1.1)

8. Primary Outcome: T 1/2 of d-Amphetamine
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 30, 48 and 72 hours post-dose
Population: PKP
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Vyvanse Alone | SPD503 + Vyvanse
Number analyzed (Participants) | 41 | 41
hours | 11.2 (1.6) | 11.2 (1.5)

ADVERSE EVENTS:
Description: Safety population consists of all subjects who received at least 1 dose of study drug and had at least 1 post-dose safety assessment.
Arm/Group | SPD503 Alone | Vyvanse Alone | SPD503 + Vyvanse
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 9/40 | 6/41 | 6/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPD503 Alone (N=40) | Vyvanse Alone (N=41) | SPD503 + Vyvanse (N=41)
Dizziness (Nervous system disorders) | 2 | 3 | 3
Dizziness Postural (Nervous system disorders) | 4 | 1 | 0
Headache (Nervous system disorders) | 3 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.